CLINICAL TRIAL: NCT06496516
Title: Transperineal Ultrasound for Assessing and Predicting Response in Hospitalized Patients with a Flare of Ulcerative Colitis
Acronym: TAPAS-UC
Status: Not yet recruiting | Type: Observational
Sponsor: Sunshine Coast Hospital and Health Service (Other)
Responsible Party: Principal Investigator, Adam Haig, Doctor, Sunshine Coast Hospital and Health Service
Other Study IDs: 109504
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Transperineal Ultrasound; Intestinal Ultrasound
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hospitalized patients with flare of ulcerative colitis

SUMMARY:
Our aim is to determine how useful transperineal ultrasound is to assess the severity of inflammation in patients with ulcerative colitis. At the moment, there is a small amount of evidence showing it may be just as good as flexible sigmoidoscopy for this purpose. It is a non-invasive test, which means if it is equivalent, it may reduce the need for invasive tests like flexible sigmoidoscopy in the future.

Patients admitted to hospital with a flare of ulcerative colitis will be invited to participate. Participants will undergo standard of care treatment and investigation. In addition to this, they will undergo a specialized non-invasive ultrasound test through the perineum (TPUS) as well as the abdomen (TA-IUS). The results from this will be compared to the current standard, flexible sigmoidoscopy. Patients will undergo repeat ultrasound and flexible sigmoidoscopy ten weeks after hospital discharge.

We aim to show that transperineal ultrasound is useful for assessing disease severity and predicting the treatment course of hospitalized patients, and may be able to replace flexible sigmoidoscopy in some circumstances.

DETAILED DESCRIPTION:
Ulcerative colitis is a chronic inflammatory disorder of the colon from which patients may experience acute disease 'flares', often requiring hospitalization. These flares may be severe and require aggressive immunomodulatory therapy to reduce morbidity and mortality. Disease severity is determined in-part by endoscopic severity, and so flexible sigmoidoscopy is indicated at admission in patients presenting with a disease flare. Not all patients respond to initial therapy, and assessing therapeutic response has traditionally been based on clinical and laboratory parameters (e.g. C-Reactive Protein, stool frequency, presence of blood). In our institution, after clinical and biochemical response, we assess for mucosal healing using flexible sigmoidoscopy, which is the treatment target set out in the STRIDE-2 guideline. This is generally performed ten weeks after admission, after stabilization on a maintenance treatment regimen and after steroids have been discontinued. Endoscopic assessment is invasive and expensive, and to optimize resource utilization there has been interest in alternative strategies to assess ulcerative colitis activity.

Intestinal ultrasound (IUS) is a well-established imaging modality and has been shown to be sensitive and specific for colonic inflammation, and correlates well with endoscopy in patients with ulcerative colitis. A major limitation of trans-abdominal IUS (TA-IUS) is that assessment of the rectum is often difficult, with suboptimal views due to the position of the rectum deep within the pelvis. As ulcerative colitis nearly always involves the rectum and may not involve the remainder of the large bowel, traditional trans-abdominal IUS may miss significant active disease. Trans-perineal ultrasound offers an easy way to visualize the rectum and could serve as a useful adjunct to TA-IUS in the assessment of ulcerative colitis response to therapy, reducing the need for endoscopic assessment at follow-up.

To date, there has been very little published data on TPUS in ulcerative colitis, though initial evidence is promising. Sagami et al. reported a strong correlation between colonoscopy and TPUS for assessment of rectal inflammation in ulcerative colitis, and reported excellent patient acceptability of TPUS, with patients expressing a preference for this modality over flexible sigmoidoscopy. These studies were conducted in a Japanese population, and there are no similar data validating the use or acceptability of TPUS in other populations.

Hypothesis:

TPUS will provide similar diagnostic accuracy when compared with flexible sigmoidoscopy in patients hospitalized with ulcerative colitis.

All patients admitted with a flare of ulcerative colitis who meet the study inclusion criteria will be offered participation in the trial as near as feasible to the time of admission. Information regarding transperineal ultrasound and the data collected during the trial will be provided in written and verbal form, and written consent will be obtained.

Data will be collected at baseline including:

* Non identifiable demographic (age, sex) and biometric (weight, body mass index)
* Laboratory values: Haemoglobin, C-Reactive protein, Albumin, ESR, Platelets
* Clinical data: Stool frequency / 24 hours, presence of blood in stool, presence of tachycardia (heart rate over 90 beats per minute, presence of fever)
* Disease and treatment data including date of diagnosis, phenotype if known, medical treatment to date, present medical treatment

These data will also be recorded at day 3 and day 5 of hospitalization (if the patient remains an inpatient), and steroid response as defined by the Oxford criteria will be documented.

All patients will undergo standard of care assessment of disease, including screening for gastrointestinal infection and a baseline flexible sigmoidoscopy as near as possible to the time of hospitalization. Disease extent and severity will be documented using the Ulcerative Colitis Index of Severity (UCEIS) score. Management will be at the discretion of the treating gastroenterologist, in line with international guidelines.

Ultrasound At the first practical opportunity after admission, all patients who consent and are enrolled will undergo transperineal ultrasound and transabdominal ultrasound. This will be carried out in a private area with an additional hospital staff member present as a chaperone during the transperineal component of the examination. Ultrasound will be carried out by an accredited intestinal ultrasound provider (staff specialist gastroenterologist) or inflammatory bowel disease fellow under supervision. Transabdominal images will be acquired using a Canon Aplio i800 with low and high frequency curvilinear or linear probe, selected at the discretion of the practitioner, depending on bowel depth and image quality. Transperineal images will be acquired using mid frequency microconvex probe.

Ultrasound image acquisition

* Unaffected segment - Two still images of each segment in longitudinal and transverse view.
* Affected segment - Cine loop of 3-10s in each segment. Colour doppler Index (CDI) cine loop 5s. Rectum - irrespective of affected or unaffected. TA-IUS - two still images in cross section. TPUS - two still images longitudinal, 3-10s cine loop in longitudinal, CDI 5s cine loop

Ultrasound data collected on each segment will include

* Bowel wall thickness
* Bowel wall doppler signal (using the modified Limberg system)
* Bowel wall stratification
* Presence of mesenteric fat echogenicity
* Presence of localized lymph nodes

Disease severity will be calculated as per the Milan criteria.

Follow up Approximately 10 weeks after admission, repeat flexible sigmoidoscopy will be performed to assess response to treatment as per our current standard practice and disease extent and severity using the UCEIS score will be documented. Laboratory data including albumin, C-Reactive protein and Haemoglobin will be recorded. In addition to this, TA-IUS and TPUS will be performed and disease severity for each of these modalities will be documented as described above.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >= 18 years old
* Presentation with a moderate or severe flare of ulcerative colitis as defined by standard clinical and laboratory criteria
* Confirmed diagnosis of ulcerative colitis or clinical history consistent with the disease
* Ability to provide informed consent and willingness to comply with study protocols

Exclusion Criteria:

* Pregnant women
* Patients with severe comorbidities for whom endoscopic assessment is contraindicated
* Patients with non-UC colitis (e.g. Crohn's colitis, ischaemic colitis)
* Patients with active perianal disease deemed by the study coordinators as severe enough to preclude the comfortable use of trans-perineal ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to the Sunshine Coast University Hospital meeting the listed eligibility criteria during the study recruitment period
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of transperineal ultrasound | At enrolment and at week 10 after hospital discharge
  The diagnostic accuracy of transperineal ultrasound when compared to the gold standard of flexible sigmoidoscopy.

SECONDARY OUTCOMES:
Additive diagnostic accuracy of transperineal ultrasound compared to transabdominal intestinal ultrasound | At enrolment and at week 10 following hospital discharge
  Additive diagnostic accuracy of transperineal ultrasound compared to transabdominal intestinal ultrasound - the absolute and relative change in diagnostic accuracy when compared to flexible sigmoidoscopy
Patient reported acceptability of transperineal ultrasound | At enrolment and at week 10 following hospital discharge
  Patient reported acceptability of transperineal ultrasound, assessed using a Likert scale, from 0 "Not at all acceptable" to 5 "Very acceptable"
Additive diagnostic accuracy of transabdominal intestinal ultrasound compared to transperineal ultrasound | At enrolment and at week 10 following hospital discharge
  Additive diagnostic accuracy of transperineal ultrasound compared to transabdominal intestinal ultrasound - the absolute and relative change in diagnostic accuracy when compared to flexible sigmoidoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Lauren S White, MBBS, Principal Investigator — Sunshine Coast Hospital and Health Service
Locations (1):
- Sunshine Coast University Hospital, Birtinya, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided
Pending site approval